CLINICAL TRIAL: NCT04500314
Title: Efficacy of Whole-body Vibration on Balance Control, Postural Stability and Mobility After Thermal Burn Injuries. Prospective Randomized Controlled Trial.
Brief Title: Efficacy of Whole-body Vibration on Balance Control, Postural Stability and Mobility After Thermal Burn Injuries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadaya Mosaad, Lecturer, department of physical therapy for surgery, Faculty of Physical Therapy , Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 182020
Record Dates: First submitted 2020-07-26; First posted 2020-08-05 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Thermal Burn

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration plus routine physical therapy (Experimental)
  Interventions: Device: whole body vibration device; Other: routine physical therapy treatment
- Routine physical therapy (Active Comparator)
  Interventions: Other: routine physical therapy treatment

INTERVENTIONS:
Device: whole body vibration device — 20 patients will receive vibration training on vibration platform (Power Plate International, Irvine, California, USA) at a frequency of 25-30 Hz and amplitude of 3-5mm, plus traditional physical therapy program 3 sessions per week for total period of 8 weeks. The total duration of the WBV training stimulus will 10 min in first week and progress gradually to 25 min in the 8th week with regular increase by 5 minutes after each 2 successive weeks
  Arms: Whole body vibration plus routine physical therapy
Other: routine physical therapy treatment — The program consists of 60 minutes supervised and individualized stretching exercise to all involved muscles followed by strengthening for affected muscles, mobilizing exercise for the joints involved to increase the joint range of motion, in addition to scar management techniques including pressure garments, inserts, and physical agent modalities , to avoid scar or contracture formation

SUMMARY:
This study will be conducted to investigate the effect of whole-body vibration device on Balance control, postural Stability and mobility after thermal burn injuries.

DETAILED DESCRIPTION:
40 patients with deep second-degree burn involving the lower limbs and trunk (TBSA: 35-40%), will be randomly assigned either into the experimental group, received whole body vibration (WBV) plus the routine physical therapy program or the control group, received the same routine physical therapy program. All treatment interventions will be applied at a frequency of three sessions per week for 8 weeks. Anteroposterior stability (APS), Medial lateral stability (MLS), Time up and go test (TUG) test, and Berg balance scale will be the outcome measures of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged between 20 and 45 years,
* Deep 2nd degree of thermal burn of lower limb and trunk with (35-40%) surface area of burn as measured by "rule of nine" method, with complete wound healing or after 6 weeks from the injury.
* Body mass index of between 17 and 35, with no history of neurological disorders or injuries to the lower extremities.

Exclusion Criteria:

* Patients with open burn wound,
* Patients diagnosed with acute rheumatoid arthritis,
* Joint replacement within the past year,
* History of traumatic spine within the past six months,
* Prosthesis,
* Recent fracture or bone disease.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Postural stability | 8 weeks of treatment
  The antero-posterior stability index (APSI) was measured for all cases before and after eight weeks of treatment. This index will be standard deviations assessing fluctuations around the zero point (horizontal) rather than around a group mean. The APSI assessed the fluctuations from the horizontal along the AP on the BSS

SECONDARY OUTCOMES:
Time up and go test | 8 weeks of treatment
  The TUG test used to measure mobility. Participants were asked to raise up from sitting in a chair to a standing position and to walk a distance of 3 m, turn around, walk back to the chair, and sit down again with their backs flush to the back of the chair and with arms resting on the arm rests. The time for participants to complete the task was measured in seconds with a stopwatch. The best, or lowest time from 3 trials, was used in the analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Faculty of physical therapy., Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after 6 month from the date of publication
Supporting Information: Study Protocol, ICF
Time Frame: After 6 month of publication.
Access Criteria: Study protocol. Informed consent form